CLINICAL TRIAL: NCT04248296
Title: Evaluate the Intestinal Microbiome in Patients With Erosive Gastroesophageal Reflux Disease and in Asymptomatic Healthy Controls
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 53677316.7.0000.0068
Record Dates: First submitted 2019-09-16; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2019-09

CONDITIONS: Gastroesophageal Reflux Disease With Esophagitis
Keywords: Gastroesophageal Reflux; intestinal microbiome
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Microbiome DNA was extracted from stool samples, and PCR amplification was performed using primers for the V4 region of the 16S rRNA gene. The amplicons were sequenced using the Ion PGM Torrent platform, and data were analyzed using QIIME™ software version 1.8 (Quantitative Insights Into Microbial Ecology).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
. In this study, we investigated intestinal microbiomes, in individuals with Gastroesophageal Reflux Disease and healthy individuals, using metagenomic techniques.

DETAILED DESCRIPTION:
Background: The pathophysiology of Gastroesophageal Reflux Disease (GERD) involves several mechanisms. Intestinal dysbiosis may influence factors involved in the pathophysiology of Gastroesophageal Reflux Disease, such as changes in gastrointestinal motor patterns and increased intraabdominal pressure due to increased fermentation of non-digestible carbohydrates. However, few studies have focused on assessment of gut microbiome in the GERD. In this study, we investigated intestinal microbiomes, in individuals with Gastroesophageal Reflux Disease and healthy individuals, using metagenomic techniques.

Methods: We performed a study comprising fecal samples of 22 adults, aged 18-60 years: 11 with erosive esophagitis (eight male and three female) and 11 healthy controls (ten male and one female). Microbiome DNA was extracted from stool samples, and polymerase chain reaction amplification was performed using primers for the V4 region of the 16S rRNA gene (16S ribosomal ribonucleic acid). The amplicons were sequenced using the Ion Torrent™ Personal Genome Machine™ platform, and data were analyzed using QIIME™ software version 1.8 (Quantitative Insights Into Microbial Ecology).

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of erosive GERD through clinical and endoscopic criteria
* who have not taken omeprazole or any other drug that changes gastric pH in the thirty days prior to the completion of diagnostic tests for GERD and other tests included in the protocol.

Exclusion Criteria:

* Use of antimicrobials or probiotics in the last three months
* Presence of severe and/or extensive atrophic gastritis confirmed histologically
* Comorbidities that could interfere with motility of the gastrointestinal tract (diabetes mellitus, previous stroke, neurological diseases)
* Use of drugs that could interfere with motility of the gastrointestinal tract or salivation (calcium channel blockers, nitrates, anticholinergics, estrogens)
* Bulky hiatal hernia (greater than or equal to 5 cm)
* Los Angeles grade C or D erosive esophagitis
* Long-distance travel in the last 3 months (outside the southeastern region of the country)
* Pregnant or breastfeeding patients
* Previous history of upper digestive tract surgery
* Obesity (body mass index equal to or greater than 30 kg / m2)
* Patient with a consumptive syndrome or malnutrition
* Tobacco use in the last 30 days / Alcohol use (more than 20 g per day, in the last 30 days)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: : We performed a study comprising fecal samples of 22 adults, aged 18-60 years: 11 with erosive esophagitis (eight male and three female) and 11 healthy controls (ten male and one female).
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Determine the microbiome | 2017-2018
  In this study, we investigated intestinal microbiomes, in individuals with Gastroesophageal Reflux Disease and healthy individuals, using metagenomic techniques. To analyze and compare different samples, we used two types of diversity indices: alpha (α) and beta (β). The relative abundance of the samples was calculated using the non-parametric Mann-Whitney test. Boxplot graphs and tables were generated to compare groups. All tests performed took into account a bidirectional α of 0.05 and a confidence interval (CI) of 95%.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clinicas da FMUSP, São Paulo, Brazil